CLINICAL TRIAL: NCT02134977
Title: Leuplin SR 11.25 mg Injection Kit Specified Drug-use Survey: "QOL Survey in Premenopausal Breast Cancer Patients"
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 265-211; JapicCTI-142513 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-04-23; First posted 2014-05-09 (Estimated); Results first posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer
Keywords: Pharmacological therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Leuprolide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Leuprorelin Acetate: Subcutaneous administration of leuprorelin acetate 11.25 mg once every 12 weeks
  Interventions: Drug: Leuprorelin Acetate

INTERVENTIONS:
Drug: Leuprorelin Acetate — Leuprorelin Acetate SR 11.25 mg Injection Kit
  Other Names: Leuplin SR 11.25 mg Injection Kit

SUMMARY:
The purpose of this survey is to examine the effect on quality of life (QOL) improvement and convenience of switching to leuprorelin acetate 3 months depot 11.25 milligram (mg) injection kit (Leuplin SR 11.25 mg injection kit) from a 4-week adjuvant therapy with a luteinizing hormone-releasing hormone analog (LH-RHa) 1 month depot over 48 weeks in premenopausal breast cancer participants in daily medical practice. Influence of condition of estrogen receptor expression on the efficacy and safety of leuprorelin acetate SR 11.25 mg injection kit was also evaluated.

DETAILED DESCRIPTION:
This survey was designed to examine the effect on QOL improvement and convenience of switching to leuprorelin acetate 3 month depot 11.25 mg injection kit (Leuplin SR 11.25 mg injection kit) from a 4-week adjuvant therapy with a LH-RHa 1 month depot over 48 weeks in premenopausal breast cancer participants in daily medical practice, as well as to evaluate the influence of condition of estrogen receptor expression on the efficacy and safety of leuprorelin acetate SR 11.25 mg injection kit .

For adults, leuprorelin acetate SR 11.25 mg injection kit (Leuplin SR 11.25 mg Injection Kit) is usually administered subcutaneously once every 12 weeks. Prior to injection, the plunger rod of the syringe is pushed upward with the needle pointed upward, allowing the entire suspension fluid contained to be transferred to the powder. The powder is then fully suspended in the fluid while ensuring that bubbles are not generated.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal breast cancer participants who meet all the following criteria are to be enrolled in the surveillance:

  1. Participants who received 4 weeks of treatment with a repository LH-RHa preparation within 1 week prior to administration of Leuplin SR 11.25 mg Injection Kit.
  2. Participants receiving Leuplin SR 11.25 mg Injection Kit as adjuvant therapy.
  3. Participants with performance status grade of 0 or 1.
  4. Participants who answered all of the questions on the "QOL check sheet (I)" at the start (Week 0) of treatment with Leuplin SR 11.25 mg Injection Kit.

Exclusion Criteria:

* Participants who meet any of the following criteria are to be excluded from the surveillance:

  1. Participants with a history of hypersensitivity to ingredient(s) in Leuplin SR 11.25 mg Injection Kit or synthetic derivatives of luteinizing hormone-releasing hormone (LH-RH) or LH-RH.
  2. Pregnant women, possibly pregnant women, and nursing mothers.
  3. Participants with advanced (T4 or M1 according to the TNM classification [General Rules for Clinical and Pathological Recording of Breast Cancer: 16th edition]) or recurrent breast cancer.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 2816 (Actual)
Dates: Start 2011-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Postmarketing Group Manager, Study Chair — Takeda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study in 351 investigative site in Japan from 21 September 2011 to 31 March 2015.
Pre-assignment Details: Participants with a historical diagnosis of premenopausal breast cancer who were switched to leuprorelin acetate sustained-release 11.25 milligram (mg) injection kit from a 4-week adjuvant therapy with a luteinizing hormone-releasing hormone analog (LH-RHa) 1 month depot preparation as a part of daily medical practice were observed.
Groups:
- Leuprorelin Acetate: Leuprorelin Acetate, 11.25 mg sustained-release injection, subcutaneously, once every 12 weeks as part of daily medical practice were observed for up to 48 weeks.
Period: Overall Study
Arm/Group | Leuprorelin Acetate
Started | 2816
Completed | 2714
Not Completed | 102
Not completed — Protocol Deviation | 102

BASELINE CHARACTERISTICS:
Population: Safety analysis set was defined as participants who received at least one dose of study medication.
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 2714
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (5.27)
Sex/Gender, Customized [Number; unit: participants]
  Female | 2714
Performance status [Number; unit: participants] — Following are Eastern Cooperative Oncology Group (ECOG) grades. 0: Fully active, perform all pre-disease activities without restriction. 1: Restricted in physically strenuous activity but ambulatory, carry out work of a light or sedentary nature. 2: Ambulatory, capable of self-care, unable to carry out any work activities, up and about greater than (>)50% of waking hours. 3: Capable of limited self-care, confined to bed or chair >50% of waking hours. 4: Completely disabled, not capable of any self-care, totally confined to bed or chair.
  participants
    Grade 0 | 2686
    Grade 1 | 28
Healthcare category [Number; unit: participants] — Participants were categorized as outpatient and inpatient.
  participants
    Outpatient | 2709
    Inpatient | 5
Presence of Complications [Number; unit: participants]
  Had no complications | 2358
  Had complications | 355
  Not determined | 1
Number of Participants with Blood Estradiol Level [Number; unit: participants]
  >=30 picogram per milliliter (pg/mL) | 219
  Less than (<) 30 pg/mL | 273
  Not measured | 2222
Blood Estradiol Level [Mean (Standard Deviation); unit: pg/mL] — Only 492 participants had data available for blood estradiol levels.
  pg/mL | 96.07 (192.148)
Blood Follicle-Stimulating Hormone (FSH) Level [Mean (Standard Deviation); unit: milli-international units/milliliter] | 15.85 (24.712)
Time from surgery to the start of treatment [Number; unit: participants]
  < 6 months | 1434
  Greater than or equal to (>=) 6 months to <1 year | 596
  >= 1 to <2 years | 401
  >= 2 years | 272
  Not determined | 11

OUTCOME MEASURES:

1. Primary Outcome: Quality of Life Questionnaire for Cancer Patients Treated With Anticancer Drugs (QOL-ACD) Total and Subscale Score at Baseline
Description: QOL-ACD score is a score used for cancer participants treated with anti-cancer drug and is a 22-item self-reported instrument assessing differences in symptom severity and health-related QOL. It includes 4 subscale domains: Daily Activities, Physical Condition, Social Activities, Mental and Psychological Status. Total and subscale scores are calculated as sum of items within each subscale: Daily Activity (items 1-6), Physical Condition (7-11), Psychological Condition (12-16), Social Attitude (17-21) and total (1-22). Face scale: 5-point score for 1 item (22). Participants answer each question on a 5-point scale (1: not at all [worst response] to 5: very much [best response]). Score range for total score is 22 to 110 and subscale score range for daily activity is 6 to 30, and for physical condition, psychological condition, and social attitude is 5 to 25. Less total/subscale scores reflect greater symptom severity and symptom impact on health-related QOL.
Time Frame: Baseline
Population: Efficacy assessment population where baseline assessment for total and subscale scores were available. Efficacy assessment population included those participants who received at least one dose of study medication and had efficacy data available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 2178
units on a scale
  Total score (n=2174) | 88.9 (11.11)
  Daily activity (n=2178) | 28.0 (3.05)
  Physical condition (n=2178) | 21.9 (2.75)
  Psychological condition (n=2178) | 19.1 (3.74)
  Social relationships (n=2177) | 16.0 (4.18)

2. Primary Outcome: QOL-ACD Total and Subscale Score at Week 12
Description: QOL-ACD score is a score used for cancer participants treated with anti-cancer drug and is a 22-item self-reported instrument assessing differences in symptom severity and health-related QOL. It includes 4 subscale domains: Daily Activities, Physical Condition, Social Activities, Mental and Psychological Status. Total and subscale scores are calculated as sum of items within each subscale: Daily Activity (items 1-6), Physical Condition (7-11), Psychological Condition (12-16), Social Attitude (17-21) and total (1-22). Face scale:5-point score for 1 item (22). Participants answer each question on a 5-point scale (1: not at all [worst response] to 5: very much [best response]). Score range for total score is 22 to 110 and subscale score range for daily activity is 6 to 30, and for physical condition, psychological condition, and social attitude is 5 to 25. Less total/subscale scores reflect greater symptom severity and symptom impact on health-related QOL.
Time Frame: Week 12
Population: Efficacy assessment population where Week 12 assessment for total and subscale scores were available. Efficacy assessment population included those participants who received at least one dose of study medication and had efficacy data available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 2035
units on a scale
  Total score (n=2031) | 88.7 (11.2)
  Daily activity (n=2034) | 27.9 (3.12)
  Physical condition (n=2034) | 21.8 (2.87)
  Psychological condition (n=2035) | 18.8 (3.81)
  Social relationships (n=2034) | 16.3 (4.15)

3. Primary Outcome: QOL-ACD Total and Subscale Score at Week 48
Description: as for outcome 1
Time Frame: Week 48
Population: Efficacy assessment population where Week 48 assessment for total and subscale scores were available. Efficacy assessment population included those participants who received at least one dose of study medication and had efficacy data available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 1662
units on a scale
  Total score (n=1658) | 89.9 (11.08)
  Daily activity (n=1662) | 28.1 (3.01)
  Physical condition (n=1662) | 22.2 (2.66)
  Psychological condition (n=1662) | 19.1 (3.71)
  Social relationships (n=1662) | 16.6 (4.10)

4. Primary Outcome: QOL-ACD Breast (QOL-ACD-B) Score at Baseline
Description: QOL-ACD-B is a part of QOL-ACD (using questionnaire items 1 to 18). QOL-ACD is a score used for cancer participants treated with anti-cancer drug and is a 22-item self-reported instrument assessing differences in symptom severity and health-related QOL. Participants answer each question on a 5-point scale (1: not at all [worst response] to 5: very much [best response]). Total score was calculated over score range 0-100 for item 1 to 18 as ((a sum of 18 items)/18-1)*25). Score for physical condition and pain was calculated over score range 0-100 for item 1 to 6 as ((a sum of 6 items)/6-1)*25)). Score for health-care and illness satisfaction was calculated over score range 0-100 for item 7 to 10 as ((a sum of 4 items)/4-1)*25)), where less scores reflect greater symptom severity and symptom impact on health-related quality of life. Means and standard deviations were calculated for the total score and score of each subscale from questionnaire items 1 to 18.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 2176
units on a scale
  Total score (n=2172) | 70.4 (13.24)
  Physical condition and pain (n=2175) | 72.3 (17.41)
  Health-care and illness satisfaction (n=2176) | 85.1 (14.12)

5. Primary Outcome: Score of QOL-ACD-B at Week 12
Description: QOL-ACD-B is a part of QOL-ACD (using questionnaire items 1 to 18). QOL-ACD is a score used for cancer participants treated with anti-cancer drug and is a 22-item self-reported instrument assessing differences in symptom severity and health-related QOL. Participants answer each question on a 5-point scale (1: not at all [worst response] to 5: very much [best response]). Total score for QOL-ACD-B is calculated as a sum of 18 items, score range: 18 to 90 where less scores reflect greater symptom severity and symptom impact on health-related quality of life. Means and standard deviations were calculated for the total score and score of each subscale from questionnaire items 1 to 18.
Time Frame: Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 2031
units on a scale
  Total score: (n=2025) | 71.0 (13.36)
  Physical condition and pain: (n=2031) | 73.1 (17.71)
  Health-care and illness satisfaction: (n=2029) | 85.2 (14.76)

6. Primary Outcome: Score of QOL-ACD-B at Week 48
Description: as for outcome 5
Time Frame: Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 1659
units on a scale
  Total score (n=1651) | 71.9 (13.50)
  Physical condition and pain (n=1659) | 74.8 (17.34)
  Healthcare and illness satisfaction (n=1656) | 84.9 (14.89)

7. Primary Outcome: Score of QOL-ACD-B Items 19, 20 and 21 at Baseline
Description: QOL-ACD-B is a part of QOL-ACD (using questionnaire items 1 to 18). For questionnaire item 19 (Did you feel inferior to your child when you interact with him/her? [due to the impact of illness and treatment]), item 20 (Did you worry about child rearing? [due to the impact of illness and treatment]), and item 21 (Do you worry about pregnancy or delivery? [due to the impact of illness and treatment]), the calculation was based on the score of each item. Each item was scored on a 5-point scale, where 1 was the worst response and 5 was the best.
Time Frame: Baseline
Population: Efficacy assessment population where baseline assessment for each item were available. Efficacy assessment population included those participants who received at least one dose of study medication and had efficacy data available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 631
units on a scale
  Item 19: (n=631) | 3.3 (1.40)
  Item 20: (n=624) | 2.9 (1.43)
  Item 21: (n=203) | 1.7 (1.01)

8. Primary Outcome: Score of QOL-ACD-B Items 19, 20 and 21 at Week 12
Description: as for outcome 7
Time Frame: Week 12
Population: Efficacy assessment population where Week 12 assessment for each item were available. Efficacy assessment population included those participants who received at least one dose of study medication and had efficacy data available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 574
units on a scale
  Item 19 (n=574) | 3.5 (1.35)
  Item 20 (n=566) | 3.3 (1.40)
  Item 21 (n=180) | 1.8 (1.09)

9. Primary Outcome: Score of QOL-ACD-B Items 19, 20 and 21 at Week 48
Description: as for outcome 7
Time Frame: Week 48
Population: Efficacy assessment population where Week 48 assessment for each item were available. Efficacy assessment population included those participants who received at least one dose of study medication and had efficacy data available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 443
units on a scale
  Item 19 (n=443) | 3.5 (1.32)
  Item 20 (n=441) | 3.2 (1.35)
  Item 21 (n=129) | 1.7 (0.97)

10. Secondary Outcome: Percentage of Participants With Reduction in Frequency of Medical Visits Due to Change in Medicinal Agents
Description: The question was with regard to the assessment of convenience associated with the changes in agents, "Did the change in agents reduce the frequency of your medical visits?" and the answers were categorized as very much reduced, somewhat reduced, unchanged. Change in medicinal agents means participants with a historical diagnosis of premenopausal breast cancer who switched to leuprorelin acetate sustained-release 11.25 mg injection kit from a 4-week adjuvant therapy with a LH-RHa 1 month depot preparation as part of daily medical practice.
Time Frame: Week 48
Population: Efficacy assessment population where Week 48 assessment for convenience assessment were available. Efficacy assessment population included those participants who received at least one dose of study medication and had efficacy data available.
Measure: Number; unit: percentage of participants
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 2396
percentage of participants
  Very much reduced | 67.7
  Somewhat reduced | 10.1
  Unchanged | 16.9
  Not determined | 5.3

11. Secondary Outcome: Percentage of Participants Who Felt Relief From Physical and Emotional Burden
Description: The question was with regard to the assessment of convenience associated with the changes in agents, "The change in agents reduced the frequency of injections by one third; for this reason, did you feel relief from physical and emotional burden?" and the answers were categorized as felt extreme relief, felt slight relief, no feeling either way, felt little relief, felt no relief.
Time Frame: Week 48
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 2396
percentage of participants
  Felt extreme relief | 34.8
  Felt slight relief | 31.6
  No feeling either way | 17.8
  Felt little relief | 7.1
  Felt no relief | 4.8
  Not determined | 3.9

12. Secondary Outcome: Percentage of Participants With Relief From Financial Burden Due to the Change in Medicinal Agents
Description: The question was with regard to the assessment of convenience associated with the changes in agents, "Did you feel relief from financial burden (example, 3 months' drug costs and transportation fee) due to the change in agents?" and the answers were categorized as felt extreme relief, felt slight relief, no feeling either way, felt little relief, felt no relief. The sum of all the categories is not 100% because of rounding error.
Time Frame: Week 48
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 2396
percentage of participants
  Felt extreme relief | 22.2
  Felt slight relief | 41.0
  No feeling either way | 21.2
  Felt little relief | 9.5
  Felt no relief | 2.4
  Not determined | 3.6

13. Secondary Outcome: Percentage of Participants Who Worried About the Effect of the Medicinal Agent
Description: The question was with regard to the assessment of convenience associated with the changes in agents, "The change in agents reduced the frequency of injections by one third; for this reason, did you worry about the effect?" and the options of the answers were not at all worried, not too worried, no thought either way, somewhat worried, and very worried.
Time Frame: Week 48
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 2396
percentage of participants
  Not at all worried | 29.7
  Not too worried | 33.8
  No thought either way | 22.4
  Somewhat worried | 9.8
  Very worried | 0.8
  Not determined | 3.5

14. Secondary Outcome: Percentage of Participants With Change in Adverse Drug Reactions Due to the Change in Medicinal Agents
Description: The question was with regard to the assessment of convenience associated with the changes in agents, "Was there a change in adverse drug reactions (e.g., menopausal-like symptoms such as hot flushes, injection-site abnormalities) due to the change in agents?" and the options of the answers were events became much less severe, events became less severe, whether or not the events became severe cannot be determined, events became slightly more severe, and events became very severe.
Time Frame: Week 48
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 2396
percentage of participants
  Events became much less severe | 1.4
  Events became less severe | 5.5
  Cannot be determined | 68.5
  Events became slightly more severe | 17.0
  Events became very severe | 3.9
  Not determined | 3.7

15. Secondary Outcome: Percentage of Participants With Change in Pain at the Time of Injection Due to the Change in Medicinal Agents
Description: The question was with regard to the assessment of convenience associated with the changes in agents, "Was there a change in pain at the time of injection due to the change in agents?" and the options of the answers were significantly relieved, slightly relieved, whether or not the pain worsened or was relieved cannot be determined, worsened slightly, and worsened significantly.
Time Frame: Week 48
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 2396
percentage of participants
  Significantly relieved | 4.7
  Slightly relieved | 10.4
  Cannot be determined | 64.9
  Worsened slightly | 14.4
  Worsened significantly | 2.1
  Not determined | 3.5

16. Secondary Outcome: Percentage of Participants With Positive Change in Agents
Description: The question was with regard to the assessment of convenience associated with the changes in agents, "Was the change in agents good?" and the options of the answers were very good, somewhat good, whether or not the change in agents was good cannot be determined, somewhat bad, very bad.
Time Frame: Week 48
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 2396
percentage of participants
  Very good | 32.0
  Somewhat good | 36.5
  Cannot be determined | 26.0
  Somewhat bad | 1.3
  Very bad | 0.5
  Not determined | 3.7

17. Secondary Outcome: Number of Participants Reporting One or More Adverse Drug Reactions
Description: Adverse drug reactions are defined as adverse events (AE) which are in the investigator's opinion of causal relationship to the study treatment. AE are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug.
Time Frame: Baseline up to Week 48
Population: Safety analysis set was defined as participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 2714
participants | 427

18. Secondary Outcome: Number of Participants Reporting One or More Serious Adverse Drug Reactions
Description: Serious adverse drug reactions are defined as serious adverse events (SAE) which are in the investigator's opinion of causal relationship to the study treatment. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The event was occurred in breast cancer female.
Time Frame: Baseline up to Week 48
Population: Safety analysis set was defined as participants who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | Leuprorelin Acetate
Number analyzed (Participants) | 2714
participants | 8

ADVERSE EVENTS:
Time Frame: Baseline up to week 48
Description: At each visit the investigator had to document any occurrence of adverse drug reactions and abnormal laboratory findings. Only adverse drug reactions were collected in this study.
Arm/Group | Leuprorelin Acetate
Serious Adverse Events (participants affected / at risk) | 8/2714
Other Adverse Events (participants affected / at risk) | 239/2714
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Leuprorelin Acetate (N=2714)
Radiation pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Metastases to lungs (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Endometriosis (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Leuprorelin Acetate (N=2714)
Hot flush (Vascular disorders) | 239

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.